CLINICAL TRIAL: NCT00454467
Title: Prospective Evaluation of the Clinical and Economic Outcomes of Total Joint Replacement: The HSS Knee Arthroplasty Cohort
Brief Title: Hospital for Special Surgery Knee Arthroplasty Cohort
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2015-093
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Knee Arthroplasty
MeSH Terms: interventions — Surveys and Questionnaires; Cost-Benefit Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Baseline Questionnaire — Patients will fill out a baseline questionnaire prior to surgery.
Procedure: Operative Data — Type of prosthesis and other operative data will be uploaded into our database.
Procedure: Intra-operative data will be collected post-operatively — Research assistants will post-operatively collect data from patient charts.
Procedure: In-hospital post-operative data will be collected — Research assistants will collect information about hospital stay from patient charts.
Procedure: Satisfaction data will be extracted from Press/Ganey and on follow-up questionnaires — Follow-up questionnaires will be mailed to participants.
Procedure: Cost Data — Cost Data will be collected via hospital billing databases.
Procedure: Follow-up questionnaires — Participants will be mailed follow-up questionnaires.

SUMMARY:
Total joint replacements are some of the most successful medical devices developed over the last fifty years. They enable millions of people to remain ambulatory and pain free, with minimal risk. In 2002, over 200,000 total hip replacements, 350,000 total knee replacements, and 25,000 total or partial shoulder replacements were performed in the United States (HCUP data). Future use will likely be even higher: it is estimated that by the year 2020, the population 65 and over in developed countries will increase by 71%. Existing studies do not provide adequate prospective data to evaluate long-term outcomes. Most health related quality of life studies in THA and TKA only report data up to twelve months post-operatively. In addition, most large studies of TKA and THA have been performed in Medicare patients. While these databases are important in providing population based data, Medicare studies do not permit any direct patient contact, and provide no information on patients under 65.

Existing studies have also investigated predictors of patient outcome at one and two years after joint arthroplasty. However, very little is known about predictors of prosthesis failure, and there are no validated clinical indicators for choosing one prosthesis model over another. Once a device is FDA approved, there is very little motivation on the part of the developer to perform complete post-marketing research, despite the importance of these data to the public health. Most existent studies are not powered to compare differences between models.

The purpose of this study is to establish a prospective cohort of HSS total knee arthroplasty.

DETAILED DESCRIPTION:
Total joint replacements are some of the most successful medical devices developed over the last fifty years. They enable millions of people to remain ambulatory and pain free, with minimal risk. In 2002, over 200,000 total hip replacements, 350,000 total knee replacements, and 25,000 total or partial shoulder replacements were performed in the United States (HCUP data). Future use will likely be even higher: it is estimated that by the year 2020, the population 65 and over in developed countries will increase by 71%. Existing studies do not provide adequate prospective data to evaluate long-term outcomes. Most health related quality of life studies in THA and TKA only report data up to twelve months post-operatively. In addition, most large studies of TKA and THA have been performed in Medicare patients. While these databases are important in providing population based data, Medicare studies do not permit any direct patient contact, and provide no information on patients under 65.

Existing studies have also investigated predictors of patient outcome at one and two years after joint arthroplasty. However, very little is known about predictors of prosthesis failure, and there are no validated clinical indicators for choosing one prosthesis model over another. Once a device is FDA approved, there is very little motivation on the part of the developer to perform complete post-marketing research, despite the importance of these data to the public health. Most existent studies are not powered to compare differences between models.

The purpose of this study is to establish a prospective cohort of HSS total knee arthroplasty.

The creation of large prospective joint arthroplasty cohorts responds directly to initiatives proposed in the NIH Consensus Development Conferences on Total Knee Replacement. This study will allow in depth analysis from the "Provider and Health Care System Perspective", (one of the important research perspectives advocated by the NIH), including surgeon, surgical technique, type of prosthesis, implantation technique and perioperative care. We will be able to evaluate all patients who receive arthroplasty surgery at HSS, as opposed to a convenience sample, and we will be able to follow patients for the life of their joint replacement. We will also be able to asses patient-level factors affecting outcomes, including medical and socio-demographic characteristics, participation in rehabilitation services, the extent of social support, and the level of patients' physical activity.

The consensus conference emphasized the importance of evaluating the use of TJA in younger patients, as these patients are underrepresented in most existing studies. For example, in one of the most rigorous existing studies of TKA, patients were followed for two years after surgery. However, three centers were needed to recruit 860 TKA patients, whose mean age was 70. By contrast, HSS alone performed over 2,000 total knee replacement surgeries in 2004, of which 41% were in patients under 65 years of age, and 28% were in patients under 60 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Undergoing total knee arthroplasty at HSS
* Pregnant women are eligible for the registry as this is a non-interventional study which only involves filling out questionnaires.

Exclusion Criteria:

* No other exclusion criteria; this is a non-interventional study which only involves filling out questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will be asking all patients undergoing total knee arthroplasty to participate.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2007-04; Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Sculco, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- See also: CERTS tools and resources — http://www.certs.hhs.gov